CLINICAL TRIAL: NCT02438982
Title: Efficacy and Safety of Rituximab to That of Calcineurin Inhibitors in Children With Steroid Dependent Nephrotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Principal Investigator, Dr. Biswanath Basu, Assistant Professor & In charge, Division of Pediatric Nephrology, Nilratan Sircar Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pednephro RCT/PM/NRSMCH-54; CTRI/2014/01/004355 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus; Calcineurin Inhibitors; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Oral Tacrolimus (Tablet form) 0.2mg/kg/day starting dose. Targeting trough level of Tacrolimus (T0) 5-7 ng/ml.
  Interventions: Drug: Tacrolimus
- Rituximab (Experimental): Two rituximab infusions will be administered once every week at standard dose (Intravenous infusion of rituximab 375mg/mt2). Circulating B cells will be measured 24 hours after rituximab administration. If >5 B cells per mm3 , it will be measured again after 1 week. If count is still >5 B cells per mm3, third & fourth doses of rituximab will be given.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Tacrolimus — Oral Tacrolimus (Tablet form) 0.2mg/kg/day starting dose. Targeting trough level of Tacrolimus (T0) 5-7 ng/ml.
  Other Names: Calcineurin inhibitor
  Arms: Tacrolimus
Drug: Rituximab — Two rituximab infusions will be administered once every week at standard dose (Intravenous infusion of rituximab 375mg/mt2). Circulating B cells will be measured 24 hours after rituximab administration. If >5 B cells per mm3, it will be measured again after 1 week. If count is still >5 B cells per mm3, third & fourth doses of rituximab will be given.
  Other Names: anti CD20 monoclonal antibody
  Arms: Rituximab

SUMMARY:
Nephrotic syndrome in children is primarily caused by minimal change disease. Majority of these patients respond well to corticosteroids. However, as many as 70% of children with nephrotic syndrome experience at least one relapse, and 30% develop a more complicated course with frequent relapses (FRNS)(≥2 relapses/ 6 months) with or without steroid dependency (SDNS)(relapse during tapering or within 2 weeks after discontinuation of corticosteroids). Repeated and prolonged courses of steroids in these children often result in long-term complications. The goal of the treatment is to reduce the rate of relapses, the cumulative dose of corticosteroids, and the incidence of serious complications. In order to minimize the side effects of steroid therapy, different steroid sparing agents such as cyclophosphamide, calcineurin inhibitors(CNI), levamisole, and mycophenolate mofetil (MMF) have been used in SDNS. Whereas CNI are usually considered the steroid sparing drug class of first choice, rituximab is increasingly used as alternative to minimize CNI toxicity. Various prospective studies suggest that Rituximab, a B cell depleting monoclonal antibody, could be a safe and effective alternative to steroid or immunosuppressants to achieve and maintain remission in this population.Single rituximab course have been shown to be efficacious for 6 to 12 months and the side effect profile observed to date is very benign. Studies comparing the usefulness of these agents are lacking. In our proposed randomized controlled trial, the investigators want to compare the efficacy and safety of CNI to that of Rituximab in treating children with SDNS.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 16 years with SDNS
* Minimal Change disease/FSGS/MesPGN/ as per Kidney Biopsy report.
* Estimated glomerular filtration rate (eGFR) >80 ml/min per 1.73 m2 at study entry.
* Remission at study entry (trace or nil proteinuria, as determined by the dipstick test or <100 mg/dl for at least 3 days).
* Not received any steroid sparing agent previously.
* Parents willing to give informed written consent.
* Ability to swallow tablet

Exclusion Criteria:

* Known etiology (e.g., lupus erythematosus, IgA nephropathy, amyloidosis, malignancy, other secondary forms of NS)
* Patients with severe leucopenia (leucocytes <3.0× 1000 cells/mm3), severe anemia (haemoglobin <8.9 g/dl), thrombocytopenia (platelet <100.0 × 1000 cells/mm3) or deranged liver function tests (AST or ALT to >50 IU/L ) at enrolment.
* Known active chronic infection (tuberculosis, HIV, hepatitis B or C) Live vaccination within 1 mo

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
12-month relapse-free survival | 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Biswanath Basu, Principal Investigator — Assistant Professor
Locations (1):
- NRS Medical College & Hospital, Kolkata, West Bengal, India

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Basu B, Sander A, Roy B, Preussler S, Barua S, Mahapatra TKS, Schaefer F. Efficacy of Rituximab vs Tacrolimus in Pediatric Corticosteroid-Dependent Nephrotic Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2018 Aug 1;172(8):757-764. doi: 10.1001/jamapediatrics.2018.1323. PMID 29913001